CLINICAL TRIAL: NCT02052323
Title: Study to Determine the Efficacy of Artesunate-mefloquine Combination Therapy for the Treatment of Uncomplicated P. Falciparum Malaria in Thailand
Brief Title: Harmonized AS/MQ Efficacy Study - Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Global Emerging Infections Surveillance and Response System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR2017
Record Dates: First submitted 2014-01-07; First posted 2014-02-03 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Malaria
Keywords: P.f Malaria, Artemisinin resistance, ACT treatment failure
MeSH Terms: conditions — Malaria | interventions — Artesunate; Mefloquine; Methaqualone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- artesunate/mefloquine (AS/MQ) (Experimental): The antimalarial drug regimen being evaluated is: artesunate (AS) 4mg/kg by mouth once daily at 0, 24 and 48 hours; plus mefloquine (MQ) 15mg/kg by mouth once at 72 hours, and 10mg/kg once by mouth at 84-96 hours; plus primaquine (PQ) 0.5mg/kg single dose by mouth at 84-96 hours
  Interventions: Drug: Artesunate/mefloquine (AS/MQ)

INTERVENTIONS:
Drug: Artesunate/mefloquine (AS/MQ) — * artesunate (AS) 4mg/kg by mouth once daily at 0, 24 and 48 hours
  * mefloquine (MQ) 15mg/kg by mouth once at 72 hours, and 10mg/kg once by mouth at 84-96 hours
  * primaquine (PQ) 0.5mg/kg single dose by mouth at 84-96 hours
  Other Names: Mequin

SUMMARY:
The purposes of this study is to determine parasitological clearance rates by microscopy for the 72-hour period after first artesunate dose in subjects with uncomplicated P. falciparum malaria.

DETAILED DESCRIPTION:
Project Summary

Objectives

Primary Objective

1. To determine parasitological clearance rates by microscopy for the 72-hour period after first artesunate dose in subjects with uncomplicated P. falciparum malaria

Secondary Objectives

2.1. To describe clinical and parasitological outcomes for subjects with uncomplicated P. falciparum malaria treated with AS-MQ administered sequentially.

2.2. To measure the gametocyte carriage rate in subjects with uncomplicated malaria before and after treatment.

2.3. To monitor drug levels associated with artesunate-mefloquine treatment failure.

2.4. To determine in vitro drug sensitivity profiles for fresh parasites from malaria-infected subjects prior to artesunate-mefloquine treatment and at the time of parasite recurrence.

2.5. To identify specific genetic determinants of artemisinin resistance derived from parasite populations.

2.6. To correlate clinical outcomes from the in vivo study with in vitro antimalarial drug sensitivity responses and molecular genotyping.

2.7. To compare P. falciparum malaria artemisinin resistance genotypes at three sites in three continents, using clinical and parasitological outcomes, in vitro drug sensitivity profiles, and molecular markers generated using harmonized methodologies.

2.8. To determine the contribution of host immunity to parasitological and clinical outcomes.

2.9. To create a catalog of parasite samples closely correlated to clinical datasets to longitudinally track resistance trends.

Subject Population

Subjects aged 5-65 years, who meet study entry criteria will be drawn from the local community.

Study Site

The study will be based at the Kwai River Christian Hospital (KRCH) in Sangklaburi District, Kanchanaburi Province, Thailand, which is located about 360km northwest of Bangkok near the Thailand-Myanmar border. Additional sites in Thailand, including in Sai Yok District, Kanchanaburi Province, may be added if enrolment at Sangklaburi is insufficient.

Number of Subjects

Up to 100 subjects will be enrolled to ensure a minimum of 59 subjects complete all study activities. This will allow for 40% subjects dropping out or being otherwise unevaluable. Up to 200 subjects may be screened to achieve the required number of evaluable subjects. A subject is considered evaluable at 72 hours from the commencement of artesunate treatment or once asexual parasites have been cleared from peripheral blood based on microscopy, whichever is longer.

Treatment

The antimalarial drug regimen being evaluated is: artesunate (AS) 4mg/kg by mouth once daily at 0, 24 and 48 hours; plus mefloquine (MQ) 15mg/kg by mouth once at 72 hours, and 10mg/kg once by mouth at 84-96 hours; plus primaquine (PQ) 0.5mg/kg single dose by mouth at 84-96 hours.

Study Design and Methodology

This is an open-label, single-arm evaluation of AS-MQ combination for the treatment of uncomplicated P. falciparum malaria. Subjects will remain as in-patients until completion of antimalarial treatment and will then be followed up weekly to 42 days.

Study Endpoints

Primary Endpoint

1. Parasite clearance rate as defined by the slope of the linear portion of the logarithm parasite clearance curve using microscopy to determine parasitemia

Secondary Endpoints

2.1. A description of the clinical and parasitological features of uncomplicated malaria in this setting (composite endpoint), including:

* Parasite clearance rate during the first 72 hours after artesunate administration as defined by the slope of the linear portion of the logarithm parasite clearance curve using qPCR to determine parasitemia
* Parasite reduction ratios at 24 and 48 hours assessed by microscopy and qPCR
* Time for parasite count to fall to 50%, 90%, 99% and 100% of initial parasite density
* Fever clearance time (i.e. the time taken for temperature to fall below 38.0˚C (tympanic method) or below 37.5˚C (axillary method) and remain there for at least 24 hours)
* 42-day PCR-adjusted treatment efficacy using World Health Organization classification of outcome.

2.2. Gametocyte carriage rates assessed in person weeks (up to 42 days) 2.3. Plasma levels of AS, DHA and MQ at selected time points 2.4. In vitro IC50, IC90, IC99 P. falciparum responses to a panel of antimalarial drugs, including dihydroartemisinin (DHA) and mefloquine.

2.5. Parasite molecular markers of drug resistance as determined by GWAS, SNP analysis and other genotyping methodologies 2.6. A detailed characterization of drug-resistant malaria using integrated endpoints above, including clinical, in vitro and molecular 2.7. Comparison of clinical and parasitological outcomes and in vitro and molecular features of parasites between harmonized sites in Kenya and Peru.

2.8. Identification of host factors that correlate with slow parasite clearance and other clinical outcomes 2.9. Creation of a well-characterised catalog of malaria parasites for future research

ELIGIBILITY:
Inclusion Criteria:

* Thai or non-Thai, otherwise healthy, male or female, aged from 5 years to 65 years inclusive
* Acute uncomplicated P. falciparum malaria monoinfection, confirmed by positive blood smear
* Asexual P. falciparum parasitaemia of 1,000 to 200,000 parasites/µL, confirmed on a thin or thick blood film
* Fever defined as ≥ 38.0°C tympanic temperature (or equivalent) or a history of fever within the last 24 hours
* Willingness to participate in the study as evidenced by written informed consent from the subject or parent/guardian (for children), and by assent (for children)

Exclusion criteria:

* Severe malaria as defined by WHO criteria (reference WHO 2012)
* Inability to eat or drink, inability to tolerate oral antimalarial medication, recent history of seizures (one or more in the previous 24 hours), altered level of consciousness, inability to sit or stand
* Mixed species asexual stage malaria infection as determined by microscopy
* Recent antimalarial treatment, defined as a clear history of any antimalarial medication taken within the previous 7 days; or a clear history of mefloquine within previous 4 weeks
* History of splenectomy
* Pregnancy or nursing mother
* Known hypersensitivity to artesunate, mefloquine or primaquine
* PI determines that it is in the best interests of the subject not to participate in the trial

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Parasite clearance rate | one year
  Parasite clearance rate as defined by the slope of the linear portion of the logarithm parasite clearance curve using microscopy to determine parasitemia

SECONDARY OUTCOMES:
Number of patients with prolonged parasite clearance times, adequate drug levels and positive molecular markers of parasite resistance. | one year
  * Parasite clearance rate during the first 72 hours after artesunate administration as defined by the slope of the linear portion of the logarithm parasite clearance curve using qPCR
  * Parasite reduction ratios at 24 and 48 hours assessed by microscopy and qPCR
  * Time for parasite count to fall to 50%, 90%, 99% and 100% of initial parasite density
  * Fever clearance time
  * 42-day PCR-adjusted treatment efficacy
  * Gametocyte carriage rates
  * Plasma levels of AS, DHA and MQ at selected time points
  * In vitro IC50, IC90, IC99 P. falciparum responses to a panel of antimalarial drugs, including dihydroartemisinin (DHA) and mefloquine
  * Parasite molecular markers of drug resistance as determined by GWAS, SNP analysis and other genotyping methodologies
  * A detailed characterization of drug-resistant malaria using integrated endpoints above, including clinical, in vitro and molecular

OTHER OUTCOMES:
Numbers of patients with features suggestive of antimalarial drug resistance in Thailand with partner sites in Kenya and Peru. | One year
  * Comparison of clinical and parasitological outcomes and in vitro and molecular features of parasites between harmonized sites in Kenya and Peru
  * Identification of host factors that correlate with slow parasite clearance and other clinical outcomes
  * Creation of a well-characterised catalog of malaria parasites for future research

CONTACTS AND LOCATIONS:
Overall Officials: Krisada Jongsakul, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (1):
- Kwai River Christian Hospital in Sangklaburi, Thong Pha Phum, Kanchanaburi, Thailand